CLINICAL TRIAL: NCT02092623
Title: Single Incision Transvaginal Mesh (Elevate® Posterior) in Treatment of Posterior Vaginal Wall Prolapse Without Concurrent Surgery - National Prospective Multicenter Study
Brief Title: Single Incision Transvaginal Mesh in Treatment of Posterior Vaginal Wall Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Helsinki University Central Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Seija Ala-Nissilä, MD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50/180/2010; 21011 (Other: TurkuUH)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Female Genital Prolapse
Keywords: Female; Prolapse surgery with transvaginal mesh; Subjective outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transvaginal posterior mesh surgery (Other): All study patients undergo transvaginal mesh operation.
  Interventions: Device: Transvaginal posterior mesh

INTERVENTIONS:
Device: Transvaginal posterior mesh — A trocar-free fixation system with low-weight mesh
  Other Names: Elevate®Posterior

SUMMARY:
Definition: To find out complications, objective and subjective outcomes of patients with symptomatic posterior vaginal wall prolapse undergoing posterior mesh operation in nine Finnish hospitals during September 2010 and August 2013. The study hypothesis is that complications are acceptable and both objective and subjective outcomes are satisfying.

DETAILED DESCRIPTION:
The aim of this study is to investigate the safety and efficacy of Elevate®Posterior transvaginal mesh kit. Secondly the investigators want to evaluate the effect of this surgical method on non-affected anterior vaginal compartment as well as patients' outcome.

This prospective multicenter national study include patients (n=111) with symptomatic posterior vaginal wall with or without apical prolapse with stage II or more. Patients were recruited at four university hospitals and five central hospitals in Finland between September 2010 and August 2013. The study protocol was approved by the Ethics Committees in participating hospitals and all attending patients gave written consent after oral and written counseling. Baseline evaluation include standardized gynecological examination in supine position using the POP-Q system. Detailed information on patients' characteristics and medical history is gathered, focusing on especially gynecological issues. Patients fill in Pelvic Floor Distress Inventory (PFDI-20) and Pelvic organ prolapse/urinary Incontinence Sexual Questionnaire (PISQ-12).

The operations are performed by qualified surgeons (n=9) familiar with transvaginal mesh surgery. Intraoperative data is collected and immediate postoperative problems are registered.

The first follow-up visit take place at three months postoperatively. Gynecological examination with POP-Q measurements are performed and complications documented. As preoperatively, PFDI-20 and PISQ-12 questionnaires are filled in by the patients.

The second visit take place at one year postoperatively. Gynecological examination with POP-Q measurements are performed and possible late complications documented. PFDI-20 and PISQ-12 questionnaires are filled in again by the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic posterior vaginal wall with or without apical prolapse with stage II or more

Exclusion Criteria:

* concomitant surgery, immunosuppressive treatment of any kind, previous or forthcoming bowel operation with low anastomosis creation and previous vaginal radiation therapy

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | up to 1 year

SECONDARY OUTCOMES:
POP-Q measurement | preoperatively, 3 months and 1 year
  Objective results of the operation (vaginal anatomy)
Pelvic floor distress inventory (PFDI-20) | preoperatively, 3 months and 1 year
  Subjective outcome of the operation on pelvic floor symptoms
Pelvic organ prolapse/urinary incontinence sexual questionnaire (PISQ-12) | preoperatively, 3 months and 1 year
  Subjective outcome of the operation on sexual functioning

CONTACTS AND LOCATIONS:
Overall Officials: Mervi Haarala, MD, Study Director — Turku University Hospital
Locations (1):
- Turku University Central Hospital, Turku, Southwest Finland, Finland